CLINICAL TRIAL: NCT05352178
Title: a New Spark in Treating Oligorecurrent Prostate Cancer: Adding Systemic Treatment to Stereotactic Body Radiotherapy or Metastasectomy: Key to Long-lasting Event-free Survival?
Brief Title: Metastasis-directed Therapy for Oligorecurrent Prostate Cancer
Acronym: SPARKLE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S65935; 2022-000066-18 (EudraCT Number)
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Prostate Cancer Recurrent; Prostate Cancer Metastatic; Metastatic Cancer; Oligometastatic Disease; Oligometastasis; Hormone Sensitive Prostate Cancer
Keywords: Androgen deprivation therapy; Androgen receptor targeted agent; Stereotactic body radiation therapy; Metastasis-directed therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Radiotherapy; Radiosurgery; Metastasectomy; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Randomized, three-arm, phase III trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MDT alone (Active Comparator): Metastasis-directed therapy alone
  Interventions: Other: Radiotherapy (SBRT) and/or surgery (metastasectomy)
- MDT + 1 month of ADT (Experimental): Metastasis-directed therapy plus one month of androgen deprivation therapy (gosereline 3.6 mg sc, leuproreline 7.5 mg sc, triptoreline 3.75 mg im)
  Interventions: Other: Radiotherapy (SBRT) and/or surgery (metastasectomy); Drug: Androgen deprivation therapy
- MDT + 6 months of ADT + anzalutamide (Experimental): Metastasis-directed therapy plus 6 months of androgen deprivation therapy (gosereline 3.6 mg sc 1x/month or gosereline 10.8 mg sc or leuproreline 7.5 mg sc 1x/month or leuproreline 45 mg sc or triptoreline 3.75 mg im 1x/month or triptoreline 11.5 mg im 1x/3months or triptoreline 22.5 mg im) and enzalutamide (4 x 40 mg each day during 6 months )
  Interventions: Other: Radiotherapy (SBRT) and/or surgery (metastasectomy); Drug: Androgen deprivation therapy; Drug: Androgen receptor targeted therapy

INTERVENTIONS:
Other: Radiotherapy (SBRT) and/or surgery (metastasectomy) — Metastasis-directed therapay (surgery and/or radiotherapy) as treatment for oligorecurrent lesions
Drug: Androgen deprivation therapy — Arm B: gosereline 3.6 mg sc, leuproreline 7.5 mg sc, triptoreline 3.75 mg im Arm C: gosereline 3.6 mg sc 1x/month or gosereline 10.8 mg sc or leuproreline 7.5 mg sc 1x/month or leuproreline 45 mg sc or triptoreline 3.75 mg im 1x/month or triptoreline 11.5 mg im 1x/3months or triptoreline 22.5 mg im
  Arms: MDT + 1 month of ADT; MDT + 6 months of ADT + anzalutamide
Drug: Androgen receptor targeted therapy — Enzalutamide
  Arms: MDT + 6 months of ADT + anzalutamide

SUMMARY:
The aim is to investigate whether the addition of short-term androgen deprivation therapy (ADT) during 1 month or short-term ADT during 6 months together with an androgen receptor targeted therapy (ARTA) to metastasis-directed therapy (MDT) significantly prolongs poly-metastatic free survival (PMFS) and/or metastatic castration-refractory prostate cancer free survival (mCRPC-FS) in patients with oligorecurrent hormone sensitive prostate cancer.

DETAILED DESCRIPTION:
Metastasis-directed therapy (MDT) has broadened the therapeutic window in patients presenting with oligorecurrent prostate cancer as it postpones the initiation of palliative androgen deprivation therapy (pADT) and its substantial side-effects for several years. Also from a biological point of view, this might be beneficial as the (early) use of ADT promotes the development of the lethal castrate-resistant state, whereby metastatic progression is driven by androgen-independent pathways. Metastasis-directed therapy with stereotactic body radiotherapy (SBRT) or surgery has shown to be able to eradicate metastases with a significant advantage concerning the pADT-free survival compared to active surveillance. And the combination of SBRT with palliative systemic treatment significantly improved overall survival (OS) when compared tot systemic treatment alone.

One of the largest retrospective analyses (191 patients) on MDT for oligorecurrent prostate cancer has been conducted previously at UZ Leuven (doi: 10.3390/cancers12082271). Estimated median pADT-free survival was 66 months and estimated median mCRPC-free survival was not reached, but 83% of patients were still free of mCRPC at 10 years.

The addition of ADT to primary radiotherapy for intermediate of high risk prostate cancer or to salvage radiotherapy has shown to improve overall survival. Within the context of SBRT for oligorecurrent disease it is not yet known whether the addition of a certain period of ADT prolongs CRPC-free survival and if so, what should be the optimal duration of this ADT administration. Moreover, the addition of an androgen receptor targeted agent (ARTA) to ADT in men with metastatic hormone sensitive prostate cancer and a treated primary tumor resulted in significantly improved clinical outcomes, also in low-volume metastatic disease.

In this clinical trial the aim is to investigate whether the addition of short-term ADT during 1 month or short-term ADT during 6 months together with an ARTA to MDT significantly prolongs poly-metastatic free survival (PMFS) and/or metastatic castration-refractory prostate cancer free survival (mCRPC-FS) in patients with oligorecurrent hormone sensitive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven initial diagnosis of prostate adenocarcinoma
* Priory treated and controlled primary tumor
* Biochemical recurrence defined by prostate-specific antigen (PSA) values >0,2 ng/ml (i.e., two consecutive increases) following radical prostatectomy + postoperative radiotherapy and a PSA value of 2 ng/ml above the nadir after high-dose RT.
* Oligorecurrent disease defined as a maximum of 5 extracranial metastases in any organ, diagnosed on PSMA PET-CT or PSMA PET-MRI reported according to the E-PSMA consensus guidelines for interpretation of PSMA-PET (26). Nodal (N1) disease can be included only when accompanied by M1a-c disease, provided that the total number of spots does not exceed 5.
* Serum testosterone level within normal range.
* WHO performance 0-2
* Age >= 18 years old
* Absence of psychological, sociological or geographical condition potentially hampering compliance with study protocol.
* Patients must be presented at the multidisciplinary board meeting and the inclusion in the trial needs approval by this board.
* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* 2. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.

Exclusion Criteria:

* Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
* Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial
* Participation in an interventional Trial with an investigational medicinal product (IMP) or device
* Serum testosterone level at castration level.
* PSA rise while on active treatment (LHRH-agonist, LHRH antagonist, anti-androgen, maximal androgen blockade, oestrogen)
* Presence of poly-metastatic disease, defined as more than 5 metastatic lesions.
* Active malignancy other than prostate cancer that could potentially interfere with the interpretation of this trial.
* Previous treatments (RT, surgery) or comorbidities rendering new treatment with SBRT impossible.
* Contra indications for intake of enzalutamide (seizure or any condition that may predispose to seizure; significant cardiovascular disease within the last three months including myocardial infarction, unstable angina, congestive heart failure, ongoing arrythmias of grade > 2 or a thromboembolic event).
* Not able to understand the treatment protocol or sign informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 873 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2032-04-25 (Estimated)

PRIMARY OUTCOMES:
Poly-metastatic free survival (PMFS) | up to 5 years after MDT
  from the last day of MDT until the first day of poly-progression which is defined as the detection > 5 new lesions at PSMA PET-CT or PSMA PET-MRI (+/- combined with MRI if needed to improve diagnostic accuracy). In case of poly-progression, pADT will be considered the standard-of-care. Other indications to start pADT are local progression of an irradiated site and/or or clinical symptoms caused by local progression. In all cases, the initiation of pADT will only be carried out after approval of the multidisciplinary tumor board. Any decision to start with pADT will be reported with date and specific reason. If recurrence occurs in 5 lesions or less a new MDT is proposed if technically feasible.

SECONDARY OUTCOMES:
Metastatic castration-refractory prostate cancer free survival (mCRPC-FS) | up to 5 years after MDT
  mCRPC-FS will be calculated from the last day of MDT until the first day of diagnosis of castration-resistant prostate cancer (CRPC). CRPC is defined according to the contemporary EAU-guidelines as the time to biochemical and/or clinical progression at castrate testosterone levels (< 50 ng/dl). Biochemical progression is defined as three consecutive PSA rises (1 week interval), of which at least 2 rises with a PSA level of > 2 ng/ml and a rise of 50% above the nadir PSA level
Biochemical progression-free survival (bPFS) | up to 5 years after MDT
  bPFS will be calculated from the last day of MDT until the first day of biochemical relapse (BcR). BcR is defined as three consecutive PSA rises (1 week interval), of which at least 2 rises with a PSA level of > 2 ng/ml and a rise of 50% above the nadir PSA level.
Clinical progression free survival (cPFS) | up to 5 years after MDT
  cPFS will be calculated from the last day of MDT until the first day of progression (local, nodal or metastatic) on PSMA PET-CT or PSMA PET-MRI. Imaging is performed in case of BcR, defined as above. Progression on PSMA PET-CT or PSMA PET-MRI will be defined as in the consensus statements on PSMA PET-CT or PSMA PET-MRI response assessment criteria in prostate cancer:
  * the appearance of 2 or more new PSMA PET-CT or PSMA PET-MRI lesions or increase of uptake or tumor PET volume of at least 30%.
  * OR the appearance of 1 new lesion with a high suspicion on PSMA PET-CT or PSMA PET-MRI
Cancer Specific Survival (CSS) | up to 10 years after MDT
  Cancer specific survival (CSS) will be calculated from last day of treatment until PCa death.
Overall Survival (OS) | up to 10 years after MDT
  Overall survival (OS) will be calculated from last day of treatment until death from any cause.
Acute and late toxicity scoring | up to 5 years after MDT
  Acute and late toxicity as a result of radiotherapy will be scores using the Common Toxicity Criteria Version 5.0 (30).
Quality of life (QOL) | up to 5 years after MDT
  Quality of life scoring using the EORTC QLQ-C30 supplement with QLQ-PR25. We will assess the quality-of-life-years with the EuroQOL classification system (EQ-5D-5L). Assessments are planned at baseline, last day of treatment, and during follow-up consultation at month M1, M3, M6, M12 and M24

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rans K, Charlien B, Filip A, Olivier H, Julie DH, Cederic D, Herlinde D, Benedikt E, Karolien G, Annouschka L, Nick L, Kenneth P, Carl S, Koen S, Hans V, Ben V, Steven J, Gert M. SPARKLE: a new spark in treating oligorecurrent prostate cancer: adding systemic treatment to stereotactic body radiotherapy or metastasectomy: key to long-lasting event-free survival? BMC Cancer. 2022 Dec 12;22(1):1294. doi: 10.1186/s12885-022-10374-0. PMID 36503429